CLINICAL TRIAL: NCT03949491
Title: Free Flap Breast Reconstruction Using Virtual Surgical Planning and 3-D Modeling
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator left the institution.
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE6118
Record Dates: First submitted 2019-04-30; First posted 2019-05-14 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Breast Reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 3-D virtual planning and medical modeling of breast (Experimental): 3-D virtual planning and medical modeling in breast cancer patients undergoing breast reconstruction.
  * Preoperative CT-Angiogram of the abdominal wall
  * Volumetric analysis preformed
  * 3D printed models made
  * Pre operative BREAST-Questionnaires given
  * Free tissue transfer performed: Operative/Dissection Time Recorded
  * Flap/Abdominal donor site complications recorded
  * Standard Digital Photography and Harris Scoring
  * BREAST-Questionnaires given at 3, 6 months
  Interventions: Procedure: 3D medical models

INTERVENTIONS:
Procedure: 3D medical models — Using 3D medical models of the abdomen, a virtual plan will assist reconstruction to clearly define and 3D model the normal and aberrant vascular anatomy of the donor site in order to decrease both operative time and dissection time. This will also allow for the proposal of incision lines to match the corresponding volumetric analysis of the transposed tissue in order to facilitate the creation of a patient specific tailored flap, which will improve the aesthetic outcomes, decrease donor site complications and improve patient satisfaction

SUMMARY:
The purpose of this study is to determine if 3D modeling and Virtual Planning Surgery can improve the clinical outcome with patient who have a mastectomy requiring breast reconstruction.

DETAILED DESCRIPTION:
Primary objective: Using 3D medical models of the abdomen, a virtual plan will assist reconstruction to clearly define and 3D model the normal and aberrant vascular anatomy of the donor site in order to decrease dissection time and secondary perioperative complications including fat necrosis and donor site complications.

Secondary objective: To propose incision lines to match the corresponding volumetric analysis of the transposed tissue in order to facilitate the creation of a patient specific tailored flap, which will improve the aesthetic outcomes.

This is a single-armed, prospective study to determine the feasibility of using 3-D virtual planning and medical modeling in breast cancer patients undergoing breast reconstruction

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed breast caner undergoing delayed or immediate breast reconstruction.
* Performance statusECOG Performance status ≤ 2
* Subjects must have normal organ and marrow function as defined below:
* Hemoglobin ≥ 10.0 g/dl
* Leukocytes ≥ 3,000/mcL
* Absolute neutrophil count ≥ 1,500/mcL
* Platelet count ≥ 100,000/mcL
* Total bilirubin within normal institutional limits
* AST (SGOT) ≤ 2.5 X institutional upper limit of normal
* ALT (SGPT) ≤ 2.5 X institutional upper limit of normal
* Serum Creatinine within normal institutional limits
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Subjects receiving any prior abdominoplasty or abdominal liposuction, or patient that plan on undergoing radiation therapy after reconstruction.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to IV contrast.
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Pregnant or breastfeeding women are excluded from this study because IV contrast and CT scans have the potential for teratogenic or abortifacient effects. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with breast cancer, breastfeeding should be discontinued.
* Unsuitable donor site volume or vasculature based on pre-operative imaging or physical exam.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Mean operative time | Up to 6 months after reconstruction
  Mean operative time using 3D medical models of the abdomen to create a virtual plan to assist reconstruction.
Mean dissection time | Up to 6 months after reconstruction
  Mean dissection time using 3D medical models of the abdomen to create a virtual plan to assist reconstruction.

SECONDARY OUTCOMES:
Aesthetic outcomes as measured by the Harris scale | Up to 1 year after reconstruction
  Aesthetic outcomes as measured by the Harris scale, which ranges from 1-4, with higher scores indicating worse outcomes.
Donor site complications | Up to 1 year after reconstruction
  Number of donor site complications will be reported
Incidence of fat necrosis as measured by a grading system | 1 week, 2 weeks, 6 weeks, 3 months, and 6 months post reconstruction.
  Incidence of fat necrosis will be measured in the postoperative period using a classification system. Grade I necrosis will be defined as minimal requiring no surgical intervention; Grade II necrosis will be minor with some aesthetic defect requiring primary excision and closure; Grade III necrosis will be defined as requiring secondary procedures after excision to achieve satisfactory cosmesis; Grade IV necrosis will involve a necrosectomy requiring a either a completely new flap or at least a second flap to address such problems; Grade V necrosis will be defined as complete flap failure 5.
  Higher grade of fat necrosis is worse.
Patient satisfaction as measured by BREAST-Q scores | Up to 1 year after reconstruction
  Patient satisfaction as measured by BREAST-Q scores which ranges from 4-16, with higher scores indicating more satisfaction with breasts.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Ghaznavi, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: at the conclusion of study and for 5 years
Access Criteria: data requestor will need to sign a data access agreement.
URL: http://redcap.ccf.org